CLINICAL TRIAL: NCT00556842
Title: Hip Fracture Evaluation With Alternatives of Total Hip Arthroplasty Versus Hemi-Arthroplasty: A Multi-Centre Randomized Trial Comparing Total Hip Arthroplasty and Hemi-Arthroplasty on Secondary Procedures and Quality of Life in Patients With Displaced Femoral Neck Fractures
Brief Title: Comparing Total Hip Arthroplasty and Hemi-Arthroplasty on Secondary Procedures and Quality of Life in Adults With Displaced Hip Fractures
Acronym: HEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Hamilton Health Sciences Corporation (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Sophies Minde Ortopedi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UM1AR063386-01 (NIH); UM1AR063386 (NIH); 1R01AR055130-01A1 (NIH); MOP 126188 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2019-11

CONDITIONS: Hip Fractures; Femoral Neck Fractures
Keywords: Hemi-Arthroplasty; Total Hip Arthroplasty
MeSH Terms: conditions — Hip Fractures; Femoral Neck Fractures | interventions — Arthroplasty, Replacement, Hip; Hemiarthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants will undergo total hip arthroplasty.
  Interventions: Device: Total hip arthroplasty
- 2 (Active Comparator): Participants will undergo hemi-arthroplasty.
  Interventions: Device: Hemi-arthroplasty

INTERVENTIONS:
Device: Total hip arthroplasty — Proscribed approaches will include minimally invasive total hip arthroplasty (i.e., two incision approaches) and hinged prostheses or capture cups. Other surgical approach aspects, the use of cemented components, the implant manufacturer, and femoral head size will not be standardized. Surgeons will use the manufacturers' specific implant guidelines for insertion.
  Other Names: THA
  Arms: 1
Device: Hemi-arthroplasty — Surgeons will use modern implants for hemi-arthroplasty, excluding non-modular, non-canal filling unipolar implants such as Moore's and Thompson's prostheses. The choice of modular unipolar versus bipolar hemi-arthroplasty will not be standardized. Whether implants are inserted with cement or a press-fit design will also not be standardized. Surgeons will use the manufacturers' specific implant guidelines for insertion.
  Other Names: HA
  Arms: 2

SUMMARY:
Each year, hip fracture, an injury that can impair independence and quality of life, occurs in about 280,000 Americans and 36,000 Canadians. By the year 2040, the annual healthcare costs associated with hip fractures are expected to reach $9.8 billion in the United States and $650 million in Canada. It is important to have in place optimal practice guidelines for the surgical handling of this injury. One type of hip fracture, called a displaced femoral neck fracture, is often treated with a hip replacement surgery. Patients undergoing a hip replacement may receive either a total hip replacement, in which the head of the femur and the hip joint socket are replaced, or a partial hip replacement, in which only the head of the femur is replaced. This study will compare the two different hip replacement procedures to determine which one results in better outcomes after surgery in adults aged 50 and older.

DETAILED DESCRIPTION:
One type of hip fracture, called a femoral neck fracture, involves a break in the narrow part of the femur bone where the head of the femur is joined to the main shaft. The break can be either undisplaced, which involves very little separation at the fracture site, or displaced, in which there is substantial separation. For displaced fractures, surgeons usually choose between internal fixation and hip arthroplasty, which is also known as hip replacement.

Patients receiving hip arthroplasty may undergo either a total hip arthroplasty or a hemi-arthroplasty. Which surgical method is best for the patient is unknown. Advocates of total hip replacement claim better improvements in patient function and quality of life. On the other hand, advocates of hemi-arthroplasty, which include most orthopaedic surgeons, claim reduced rates of dislocation and deep vein thrombosis, shorter operating times, less blood loss, and a technically less demanding surgical procedure. This study will compare total hip arthroplasty and hemi-arthroplasty on rates of revision surgery 2 years after patients aged 50 and older sustain femoral neck fractures and undergo surgery. The study will also compare the impact of the two different surgical procedures on function, quality of life, and post-surgical complications. Results from this study may impact current orthopaedic practice.

Participation in this study will last 2 years. Before surgery, participants will complete a baseline assessment that will include x-rays, a medical history review, and a physical examination. Participants will then be randomly assigned to undergo either total hip arthroplasty or hemi-arthroplasty to repair their hip fractures. All surgeons will need to meet certain criteria to partake in the study and will have expertise in whichever surgical procedure they are performing. Surgeons will also follow the manufacturers' implant guidelines during surgery. Specific aspects of both the preoperative and post-operative care, such as weight bearing status, the prevention of thromboembolic disease, and the use of antibiotics and calcium supplementation, will be standardized for all participants. Within 2 days of under going surgery, x-rays will be performed again.

Follow-up assessments will be completed either by phone or in-person at the hospital or clinic. They will occur 1 and 10 weeks after surgery and 6, 9, 12, 18, and 24 months after surgery. All assessments will include questionnaires and interviews on health status, hip function, pain, functional mobility, and revision surgery. Some of the in-person assessments will also include x-rays.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women aged 50 years and old (with no upper age limit)
* Fracture of the femoral neck, as confirmed with either anteroposterior or lateral hip radiographs, computed tomography, or magnetic resonance imaging (MRI)
* Displaced fracture that is not, in the judgment of the attending surgeon, optimally managed by reduction and internal fixation
* Operative treatment is planned within 72 hours of the patient being medically cleared for surgery
* Patient was ambulatory prior to the fracture, though they may have used an aid such as a cane or a walker
* Anticipated medical optimization for arthroplasty of the hip
* Provision of informed consent by patient or proxy
* Low energy fracture (defined as a fall from standing height), with no other trauma
* Assurance from site that surgeons with expertise in both total hip arthroplasty and hemi-arthroplasty are available to perform surgery (Note: Surgeons do not need to be experts in both techniques)

Exclusion Criteria:

* Not suitable for hemi-arthroplasty (i.e., inflammatory arthritis, rheumatoid arthritis, pathologic fractures (secondary to cancer), or severe osteoarthritis of the hip)
* Associated major injuries of the lower extremity (e.g., ipsilateral or contralateral fractures of the foot, ankle, tibia, fibula, knee, or femur; dislocations of the ankle, knee, or hip; or femoral head defects or fracture)
* Retained hardware around the affected hip that will interfere with arthroplasty
* Infection around the hip (soft tissue or bone)
* Bone metabolism disorder except osteoporosis (e.g., Paget's disease, renal osteodystrophy, osteomalacia)
* Patients with a previous history of frank dementia that would interfere with the assessment of primary outcome (e.g., secondary procedures at 2 years).
* Likely problems, in the judgment of the investigators, with maintaining follow-up (e.g., no fixed address, plans to move out of town in the next year, or intellectually challenged and without adequate family support)
* Enrolled in another ongoing drug or surgical intervention trial
* Patients whose fracture occurred as a result of violence.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1495 (Actual)
Dates: Start 2009-03; Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Bhandari, MD PhD FRCSC, Principal Investigator — McMaster University; Thomas A. Eihnorn, MD, Principal Investigator — Boston University
Locations (2):
- New York University Medical Center, New York, New York, United States
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hebert-Davies J, Laflamme GY, Rouleau D; HEALTH and FAITH investigators. Bias towards dementia: are hip fracture trials excluding too many patients? A systematic review. Injury. 2012 Dec;43(12):1978-84. doi: 10.1016/j.injury.2012.08.061. Epub 2012 Sep 19. PMID 22999009
- [Background] Burgers PT, Van Geene AR, Van den Bekerom MP, Van Lieshout EM, Blom B, Aleem IS, Bhandari M, Poolman RW. Total hip arthroplasty versus hemiarthroplasty for displaced femoral neck fractures in the healthy elderly: a meta-analysis and systematic review of randomized trials. Int Orthop. 2012 Aug;36(8):1549-60. doi: 10.1007/s00264-012-1569-7. Epub 2012 May 24. PMID 22623062
- [Background] Burgers PT, Hoogendoorn M, Van Woensel EA, Poolman RW, Bhandari M, Patka P, Van Lieshout EM; HEALTH Trial Investigators. Total medical costs of treating femoral neck fracture patients with hemi- or total hip arthroplasty: a cost analysis of a multicenter prospective study. Osteoporos Int. 2016 Jun;27(6):1999-2008. doi: 10.1007/s00198-016-3484-z. Epub 2016 Jan 28. PMID 26821137
- [Background] Bhandari M, Devereaux PJ, Einhorn TA, Thabane L, Schemitsch EH, Koval KJ, Frihagen F, Poolman RW, Tetsworth K, Guerra-Farfan E, Madden K, Sprague S, Guyatt G; HEALTH Investigators. Hip fracture evaluation with alternatives of total hip arthroplasty versus hemiarthroplasty (HEALTH): protocol for a multicentre randomised trial. BMJ Open. 2015 Feb 13;5(2):e006263. doi: 10.1136/bmjopen-2014-006263. PMID 25681312
- [Background] Burgers PT, Poolman RW, Van Bakel TM, Tuinebreijer WE, Zielinski SM, Bhandari M, Patka P, Van Lieshout EM; HEALTH and FAITH Trial Investigators. Reliability, validity, and responsiveness of the Western Ontario and McMaster Universities Osteoarthritis Index for elderly patients with a femoral neck fracture. J Bone Joint Surg Am. 2015 May 6;97(9):751-7. doi: 10.2106/JBJS.N.00542. PMID 25948522
- [Derived] HEALTH Investigators; Bhandari M, Einhorn TA, Guyatt G, Schemitsch EH, Zura RD, Sprague S, Frihagen F, Guerra-Farfan E, Kleinlugtenbelt YV, Poolman RW, Rangan A, Bzovsky S, Heels-Ansdell D, Thabane L, Walter SD, Devereaux PJ. Total Hip Arthroplasty or Hemiarthroplasty for Hip Fracture. N Engl J Med. 2019 Dec 5;381(23):2199-2208. doi: 10.1056/NEJMoa1906190. Epub 2019 Sep 26. PMID 31557429

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Hip Arthroplasty: Participants will undergo total hip arthroplasty.
  Total hip arthroplasty: Proscribed approaches will include minimally invasive total hip arthroplasty (i.e., two incision approaches) and hinged prostheses or capture cups. Other surgical approach aspects, the use of cemented components, the implant manufacturer, and femoral head size will not be standardized. Surgeons will use the manufacturers' specific implant guidelines for insertion.
- Hemi-arthroplasty: Participants will undergo hemi-arthroplasty.
  Hemi-arthroplasty: Surgeons will use modern implants for hemi-arthroplasty, excluding non-modular, non-canal filling unipolar implants such as Moore's and Thompson's prostheses. The choice of modular unipolar versus bipolar hemi-arthroplasty will not be standardized. Whether implants are inserted with cement or a press-fit design will also not be standardized. Surgeons will use the manufacturers' specific implant guidelines for insertion.
Period: Overall Study
Arm/Group | Total Hip Arthroplasty | Hemi-arthroplasty
Started | 749 | 746
Completed | 718 | 723
Not Completed | 31 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Hip Arthroplasty | Hemi-Arthroplasty | Total
Number analyzed (Participants) | 718 | 723 | 1441
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.1 (8.3) | 78.6 (8.6) | 78.8 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 510 | 499 | 1009
  Male | 208 | 224 | 432
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Native or Aboriginal | 2 | 1 | 3
  South Asian | 3 | 6 | 9
  East Asian | 7 | 7 | 14
  Hispanic or Latino | 7 | 6 | 13
  White | 683 | 684 | 1367
  Black | 12 | 15 | 27
  Middle Eastern | 1 | 1 | 2
Prefracture Living Status [Count of Participants; unit: Participants]
  Institutionalized | 30 | 27 | 57
  Not institutionalized | 688 | 696 | 1384
Prefracture Functional Status [Count of Participants; unit: Participants]
  Uses assistive device for ambulation | 187 | 182 | 369
  Able to ambulate without assistive device | 531 | 541 | 1072
Previous Surgery to Affected Hip [Count of Participants; unit: Participants] | 2 | 1 | 3
Major Coexisting Conditions [Number; unit: participants]
  Osteopenia | 28 | 30 | 58
  Osteoporosis | 114 | 110 | 224
  Lung disease | 127 | 122 | 249
  Diabetes | 135 | 145 | 280
  Ulcers or stomach disease | 49 | 67 | 116
  Kidney disease | 71 | 67 | 138
  Anemia or other blood disease | 48 | 55 | 103
  Depression | 70 | 84 | 154
  Cancer | 65 | 80 | 145
  Osteoarthritis, degenerative arthritis | 111 | 91 | 202
  Back pain | 64 | 71 | 135
  Rheumatoid arthritis | 13 | 21 | 34
  Heart disease | 247 | 249 | 496
  High blood pressure | 434 | 443 | 877

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Revision Surgery
Description: The primary outcome is any unplanned secondary procedure within 2 years of the initial joint replacement surgery.
Time Frame: Measured 2 years after original surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Total Hip Arthroplasty | Hemi-arthroplasty
Number analyzed (Participants) | 718 | 723
Participants | 57 | 60

2. Secondary Outcome: Hip Function and Pain
Description: Hip function and pain were measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), which is a self-administered questionnaire that assesses 3 dimensions of pain, disability, joint stiffness in knee and hip osteoarthritis. This questionnaire uses a Likert scale, with the responses: none, mild, moderate, severe, and extreme. A higher score indicates worse pain, stiffness, and functional limitations. The ranges are: 0-20 for pain, 0-8 for stiffness, 0-68 for physical function. The sum of the pain, stiffness, and physical function subscales provides the WOMAC total score, which ranges from 0-96.
Time Frame: Measured 2 years after original surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Total Hip Arthroplasty: WOMAC scores for the THA group at 24 months.
- Hemiarthroplasty: WOMAC scores for the HA group at 24 months.
Arm/Group | Total Hip Arthroplasty | Hemiarthroplasty
Number analyzed (Participants) | 718 | 723
units on a scale
  WOMAC total score | 14.29 (15.64) | 17.22 (16.99)
  WOMAC pain score | 1.65 (2.97) | 2.21 (3.35)
  WOMAC stiffness score | 1.05 (1.44) | 1.22 (1.63)
  WOMAC function score | 11.13 (12.34) | 13.09 (13.00)
Statistical Analysis 1: Comparison: Total Hip Arthroplasty vs Hemiarthroplasty; Using a multi-level model, the effect of THA versus HA on function (WOMAC) was estimated. We chose an alpha level of 0.01. The results below are the mean difference in score for WOMAC total at 24 months; Test type: Equivalence — Please refer to the protocol paper for details of the power calculation; Mean Difference (Final Values) = -6.37, 99% CI 2-sided [-9.18 to -3.56]
Statistical Analysis 2: Comparison: Total Hip Arthroplasty vs Hemiarthroplasty; Using a multi-level model, the effect of THA versus HA on function (WOMAC) was estimated. We chose an alpha level of 0.01. The results below are the mean difference in score for WOMAC pain at 24 months; Test type: Equivalence — Please refer to the protocol paper for details of the power calculation; Mean Difference (Final Values) = -0.93, 99% CI 2-sided [-1.42 to -0.44]
Statistical Analysis 3: Comparison: Total Hip Arthroplasty vs Hemiarthroplasty; Using a multi-level model, the effect of THA versus HA on function (WOMAC) was estimated. We chose an alpha level of 0.01. The results below are the mean difference in score for WOMAC stiffness at 24 months; Test type: Equivalence — Please refer to the protocol paper for details of the power calculation; Mean Difference (Final Values) = -0.44, 99% CI 2-sided [-0.65 to -0.23]
Statistical Analysis 4: Comparison: Total Hip Arthroplasty vs Hemiarthroplasty; Using a multi-level model, the effect of THA versus HA on function (WOMAC) was estimated. We chose an alpha level of 0.01. The results below are the mean difference in score for WOMAC function at 24 months; Test type: Equivalence — Please refer to the protocol paper for details of the power calculation; Mean Difference (Final Values) = -4.97, 99% CI 2-sided [-7.11 to -2.83]

3. Secondary Outcome: Number of Participants With Functional Mobility Problems
Description: Functional outcome measured using the Timed Up and Go (TUG) test. The TUG test is a standardized, physical test to assess balance and mobility in the participants. The participant is timed while they perform simple physical movements, such as rising from an arm chair, walking 10 feet, walking back to the chair, and sitting down. A faster time indicates that the participant has greater functional performance, while a lower score may identify participants who are at risk for increased falls in the community.
  We analyzed the TUG as a dichotomous outcome with the following categories: a) patients who complete the test in ≤12 seconds, and b) those who require >12 seconds to complete the test or were unable to complete the test. We selected 12 seconds as the cut-off because this was the threshold used by the Centers for Disease Control and Prevention. We report the number of participants in each group who required >12 seconds to complete the test or were unable to complete the test
Time Frame: Measured 2 years after original surgery
Measure: Count of Participants; unit: Participants
Groups:
- Total Hip Arthroplasty: THA Participants who took more than 12 seconds to complete the TUG test or were unable to complete the test.
- Hemiarthroplasty: HA Participants who took more than 12 seconds to complete the TUG test or were unable to complete the test.
Arm/Group | Total Hip Arthroplasty | Hemiarthroplasty
Number analyzed (Participants) | 718 | 723
Participants | 210 | 206
Statistical Analysis 1: Comparison: Total Hip Arthroplasty vs Hemiarthroplasty; Using a multi-level model, the effect of THA versus HA on mobility (TUG) was estimated. We analyzed the TUG as a dichotomous outcome with the following categories: a) patients who complete the test in ≤12 seconds, and b) those who require >12 seconds to complete the test or were unable to complete the test. We selected 12 seconds as the cut-off because this was the threshold used by the Centers for Disease Control and Prevention. The TUG was summarized using odds ratios and 99% CIs; Test type: Equivalence — Please refer to the protocol paper for details of the power calculation; Odds Ratio (OR) = 0.72, 99% CI 2-sided [0.38 to 1.36]

4. Secondary Outcome: Health-Related Quality of Life (SF-12)
Description: Health-related quality of life measured using the SF-12 Health Survey, which is a standardized instrument to measure health- related quality of life. This self-administered, 12-item questionnaire covers eight main health domains that make up the Physical and Mental Health Composite Scores (PCS & MCS). Each domain consists of one or two questions and is scored separately from 0 (lowest level) to 100 (highest level). Higher scores represent better health-related quality of life.
Time Frame: Measured 2 years after original surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Total Hip Arthroplasty: SF-12 scores for the THA group at 24 months.
- Hemiarthroplasty: SF-12 scores for the HA group at 24 months.
Arm/Group | Total Hip Arthroplasty | Hemiarthroplasty
Number analyzed (Participants) | 718 | 723
units on a scale
  SF-12 PCS | 41.89 (11.25) | 41.27 (11.34)
  SF-12 MCS | 54.03 (9.77) | 51.36 (11.83)
Statistical Analysis 1: Comparison: Total Hip Arthroplasty vs Hemiarthroplasty; Using a multi-level model, the effect of THA versus HA on quality of life (SF-12) was estimated. We chose an alpha level of 0.01. The results below are the mean difference in score for SF-12 PCS at 24 months; Test type: Equivalence — Please refer to the protocol paper for details of the power calculation; Mean Difference (Final Values) = 1.41, 99% CI 2-sided [-0.33 to 3.14]
Statistical Analysis 2: Comparison: Total Hip Arthroplasty vs Hemiarthroplasty; Using a multi-level model, the effect of THA versus HA on quality of life (SF-12) was estimated. We chose an alpha level of 0.01. The results below are the mean difference in score for SF-12 MCS at 24 months; Test type: Equivalence — Please refer to the protocol paper for details of the power calculation; Mean Difference (Final Values) = 1.34, 99% CI 2-sided [-0.38 to 3.05]

5. Secondary Outcome: Health-Related Quality of Life (EQ-5D)
Description: Health-related quality of life was measured using the EQ-5D, which is a standardized instrument that comprises of a short descriptive system questionnaire and a visual analogue scale (EQ-5D VAS).
  The questionnaire provides a simple descriptive profile of a respondent's health state. When the descriptive system profile is linked to a 'value set', a single summary index value for health status on a 0 to 1 scale is derived that can be used in economic evaluations of healthcare interventions. A health utility value of 1 indicates perfect health while a score of 0 indicates death.
  The EQ-5D VAS assesses the individual's health today on a scale from 0-100, with the 0 being 'worst imaginable state of health' and 100 being 'best imaginable state of health'.
Time Frame: Measured 2 years after original surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Total Hip Arthroplasty: EQ-5D scores for the THA group at 24 months.
- Hemiarthroplasty: EQ-5D scores for the HA group at 24 months.
Arm/Group | Total Hip Arthroplasty | Hemiarthroplasty
Number analyzed (Participants) | 718 | 723
units on a scale
  EQ-5D utility index score | 0.82 (0.19) | 0.77 (0.22)
  EQ-5D VAS score | 72.26 (18.76) | 70.84 (19.44)
Statistical Analysis 1: Comparison: Total Hip Arthroplasty vs Hemiarthroplasty; Using a multi-level model, the effect of THA versus HA on quality of life (EQ-5D) was estimated. We chose an alpha level of 0.01. The results below are the mean difference in score for EQ-5D utility index at 24 months; Test type: Equivalence — Please refer to the protocol paper for details of the power calculation; Mean Difference (Final Values) = 0.04, 99% CI 2-sided [-0.03 to 0.11]
Statistical Analysis 2: Comparison: Total Hip Arthroplasty vs Hemiarthroplasty; Using a multi-level model, the effect of THA versus HA on quality of life (EQ-5D) was estimated. We chose an alpha level of 0.01. The results below are the mean difference in score for EQ-5D VAS at 24 months; Test type: Equivalence — Please refer to the protocol paper for details of the power calculation; Mean Difference (Final Values) = 0.72, 99% CI 2-sided [-2.02 to 3.46]

6. Secondary Outcome: Complications, Including Mortality, Dislocation, Infection, Femoral Fracture, Deep Venous Thrombosis, and Prosthesis Loosening
Description: Hip-related complications including peri-prosthetic fracture, hip instability or dislocation, implant failure (loosening/subsidence and breakage), would healing problems (including superficial/deep infection, wound necrosis), soft tissue problems (e.g. pseudotumor), heterotopic ossification, abductor failure, implant wear and corrosion, osteolysis, neurovascular injury, decreased function, or pain. Measured at 1 and 10 weeks, 6, 9,12, 18, 24 months.
Time Frame: Measured 2 years after original surgery
Measure: Number; unit: participants
Arm/Group | Total Hip Arthroplasty | Hemi-arthroplasty
Number analyzed (Participants) | 718 | 723
participants
  Death | 103 | 95
  Serious adverse event | 300 | 265
  Any hip-related complication | 132 | 118

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the 24 month follow-up period.
Arm/Group | Total Hip Arthroplasty | Hemi-arthroplasty
All-Cause Mortality (participants affected / at risk) | 103/718 | 95/723
Serious Adverse Events (participants affected / at risk) | 300/718 | 265/723
Other Adverse Events (participants affected / at risk) | 132/718 | 118/723
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Hip Arthroplasty (N=718) | Hemi-arthroplasty (N=723)
Hip fracture-related serious adverse event (Musculoskeletal and connective tissue disorders) | 59 | 57
Neurologic serious adverse event (Nervous system disorders) | 28 | 26
Respiratory serious adverse event (Respiratory, thoracic and mediastinal disorders) | 42 | 37
Cardiac serious adverse event (Cardiac disorders) | 51 | 49
Renal serious adverse event (Renal and urinary disorders) | 23 | 22
Vascular serious adverse event (Vascular disorders) | 22 | 16
Other serious adverse event (Musculoskeletal and connective tissue disorders) | 201 | 177 — including: non-trial related fracture, non-trial related dislocation, other non-trial related injury, cellulitis, death, multiorgan failure, osteoporosis, sepsis, reported by site as "other"
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Hip Arthroplasty (N=718) | Hemi-arthroplasty (N=723)
Periprosthetic fracture (Musculoskeletal and connective tissue disorders) | 38 | 35
Hip instability or dislocation (Musculoskeletal and connective tissue disorders) | 34 | 17
Superficial surgical-site infection (Musculoskeletal and connective tissue disorders) | 9 | 6
Deep surgical-site infection (Musculoskeletal and connective tissue disorders) | 17 | 16
Another wound-healing problem (Musculoskeletal and connective tissue disorders) | 6 | 5
Another soft-tissue procedure (Musculoskeletal and connective tissue disorders) | 11 | 11
Clinically important heterotopic ossification (Musculoskeletal and connective tissue disorders) | 29 | 24
Abductor failure (Musculoskeletal and connective tissue disorders) | 1 | 3
Implant failure: loosening or subsidence (Musculoskeletal and connective tissue disorders) | 5 | 5
Implant failure: breakage (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain (Musculoskeletal and connective tissue disorders) | 6 | 12
Neurovascular injury: technical error (Musculoskeletal and connective tissue disorders) | 2 | 1
Other (Musculoskeletal and connective tissue disorders) | 7 | 13

LIMITATIONS AND CAVEATS:
Patients and end-point assessors were unblinded in the assessments of function. Loss to follow-up was 14.9% for the final analysis. Data on function were incomplete; 82.9% of patients completed at least one questionnaire over 24 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT00556842/SAP_000.pdf
  • Study Protocol (2014-01-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT00556842/Prot_001.pdf